CLINICAL TRIAL: NCT05164666
Title: An Open-Label, Dose Escalation, Phase 1, First-in-Human Study of TAK-103 in Adult Patients With Mesothelin-Expressing Advanced or Metastatic Solid Tumors
Brief Title: A Study of TAK-103 in Adult With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision unrelated to patient safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-103-1001; jRCT2033210463 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-11-23; First posted 2021-12-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-103, Dose Escalation (Experimental): TAK-103, Chimeric antigen receptor (CAR) (+) cells, intravenous infusion, will be administered at approximately 5 mL/min. There are 5 planned dose levels: 1x10^6, 3x10^6, 1x10^7, 1x10^8 and 5x10^8 CAR (+) cells/body. The level of dose in dose escalation will be guided by dose escalation schema based on the observed dose limiting toxicities (DLT) rate at each dose level.
  Interventions: Biological: TAK-103

INTERVENTIONS:
Biological: TAK-103 — TAK-103 intravenous infusion

SUMMARY:
In this study, people with mesothelin-expressing advanced or metastatic solid tumors will receive TAK-103 with their white blood cells. The main aims of this study are to check if the participants get any side effects from treatment with TAK-103 and to check how much TAK-103 participants can receive without getting side effects from it. Researchers can then work out the best dose of TAK-103 to give to participants in future studies.

At the first visit, the study doctor will check who can take part. For those who can take part, the study doctors will collect white blood cells from each participant. These cells are sent to the laboratory where TAK-103 is added to each participant's cells. This can take up to 4 or 5 weeks. Participants may receive specific treatments while participants are waiting for TAK-103. Then, participants will receive TAK-103 with their cells slowly through a vein (infusion). Participants will receive lower to higher doses of TAK-103. Each participant will just receive 1 dose. The study doctors will check for side effects after each different dose of TAK-103. In this way, researchers can work out the best dose of TAK-103 to give to participants in future studies.

Participants will stay in hospital for 28 days or longer for their treatment. Then, participants will visit the clinic for regular check-ups for up to 3 years.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed advanced or metastatic solid tumors who have no option with or are intolerant of standard therapies with a proven clinical benefit.
2. Mesothelin-expression (>=50% positive on viable tumor cells) must be determined on the tumor by immunohistochemistry using a validated assay, scoring and staining confirmed by the sponsor prior to leukapheresis procedures.
3. Life expectancy >=12 weeks.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Adequate organ function as confirmed by clinical laboratory values as specified below:

   1. Total bilirubin =<1.5 × the upper limit of the normal range (ULN) except in Participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll with direct bilirubin =<3 × ULN of the direct bilirubin. Elevated indirect bilirubin due to posttransfusion hemolysis is allowed
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be <3 × ULN.

      AST and ALT may be elevated up to 5 × ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in the liver.
   3. Calculated creatinine clearance >50 mL/min (Cockcroft-Gault formula).
   4. Hemoglobin must be >=9 g/dL.
   5. Neutrophil count must be >1000/mm^3.
   6. Absolute lymphocyte count must be >500/mm^3.
   7. Platelet count must be >75,000/mm^3.
6. Participants must have radiographically measurable disease as defined by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).

Exclusion Criteria

1. Active systemic infections.
2. Known hepatitis B surface antigen (HBsAg) positive, or known or suspected active hepatitis C virus (HCV) infection. Participants who have positive hepatitis B core antibody (HBcAb) or hepatitis B surface antibody (HBsAb) can be enrolled but must have an undetectable hepatitis B virus (HBV) viral load. Participants who have positive hepatitis C virus antibody (HCVAb) must have an undetectable HCV viral load.
3. Coagulation disorders, or other major medical illnesses including respiratory or immune system disease.
4. Participants with high tumor burden at the disease assessment at screening. The tumor burden is determined by the threshold set for each type of cancer.
5. Participants with current or history of interstitial lung disease.
6. Participants with current or history of significant immune-related adverse events (irAEs) related to treatment with immune checkpoint inhibitors. Patients with current or history of the following adverse events (AEs) can be enrolled after careful discussion between the investigator and sponsor: hyperglycemia/diabetes mellitus, thyroid disorder, hypopituitarism, hypoadrenocorticism, asymptomatic elevation in amylase/lipase, and Grade1 or 2 skin toxicity.
7. Participants with known cardiovascular and cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, myocardial infarction, congestive heart failure, left ventricular ejection fraction (LVEF) <45 %, impaired respiratory function, baseline oxygen saturation <93% on room air. A well-controlled atrial fibrillation would not be an exclusion whereas uncontrolled atrial fibrillation would be an exclusion.
8. Participants with any signs of lymphoma and/or leukemia.
9. Participants who are diagnosed with or treated for another malignancy within 3 years before leukapheresis procedures. Participants with non-melanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast) would be included if they were adequately treated.
10. Any disease requiring systemic steroid treatment.
11. Any prior use of cell and gene therapy(ies).
12. Treatment with any investigational products (except for cell or gene therapy) within 14 days before leukapheresis procedures or 28 days before treatment with conditioning chemotherapy/TAK-103.
13. Systemic anticancer therapy (including immuno-oncology therapies) and treatment with radiotherapy within 14 days before leukapheresis procedures or treatment with conditioning chemotherapy/TAK-103.
14. Treatment with major surgery within 28 days before leukapheresis procedures or treatment with conditioning chemotherapy/TAK-103 (minor surgical procedures such as catheter placement are not exclusionary criteria).
15. Previous treatment with any mesothelin-targeted therapy.
16. Any unresolved toxicity of Grade 3 or higher from previous anticancer therapy.
17. Participants with risk of bleeding as judged by the investigator.
18. Presence of central nervous system metastasis or other significant neurological conditions (Participant with central nervous system metastases that have been effectively treated where necessary and stable can be enrolled).
19. Participants with human immunodeficiency virus (HIV) seropositive and/or human T-cell lymphotropic virus (HTLV) seropositive.
20. Participants with a history of organ transplantation or awaiting organ transplantation.
21. Participants with severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or streptomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Up to 28 days
  Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Percentage of Participants With Treatment-emergent Adverse Event (TEAE) | Up to 1 years
  An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug.
Percentage of Participants With Adverse Events of Clinical Interest | Up to 1 years
  Adverse events of clinical interest include severe immune effector cell-associated neurotoxicity syndrome (ICANS), cytokine release syndrome (CRS), hemophagocytic lymphohistiocytosis (HLH), macrophage activation syndrome (MAS), and tumor lysis syndrome (TLS).

SECONDARY OUTCOMES:
Overall response rate (ORR) Assessed by Investigator with RECIST 1.1 | Up to 3 years
  ORR is defined as the percentage of participants whose best overall response is complete response (CR/iCR) or partial response (PR/iPR) as determined by the investigator per RECIST 1.1 and iRECIST respectively. Disease response criteria on RECIST 1.1 are following; Complete response (CR): Disappearance of all target lesions. Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
ORR Assessed by Investigator with immune RECIST (iRECIST) | Up to 3 years
  ORR is defined as the percentage of participants whose best overall response is complete response (CR/iCR) or partial response (PR/iPR) as determined by the investigator per RECIST 1.1 and iRECIST respectively. Disease response criteria on iRECIST are following; Complete Response (iCR), which describes the complete disappearance of target lesion (TL) and Non-TL. All lymph nodes must be non-pathological in size (< 10 mm in short axis diameter [SAD]). Partial Response (iPR), which occurs when the tumor load of the TL is reduced by =<30% compared to the baseline, or in the case of complete remission of the TL, when one or more, Non-TL can still be distinguished. Stable Disease (iSD), which is to be determined if the criteria of iCR or iPR are not met and no tumor progression is present.
Disease Control Rate (DCR) Assessed by Investigator with RECIST 1.1 | Up to 3 years
  DCR is defined as the proportion of patients whose best overall response is stable disease (SD/iSD) or better as determined by the investigator per RECIST 1.1 and iRECIST respectively. SD/iSD have to be maintained for at least 24 days (around 4 weeks) after the TAK-103 infusion.
DCR Assessed by Investigator with iRECIST | Up to 3 years
  DCR is defined as the proportion of patients whose best overall response is stable disease (SD/iSD) or better as determined by the investigator per RECIST 1.1 and iRECIST respectively. SD/iSD have to be maintained for at least 24 days (around 4 weeks) after the TAK-103 infusion.
Duration of Response (DOR) Assessed by Investigator with RECIST 1.1 | Up to 3 years
  DOR is defined as the time from the date of first documentation of a PR/iPR or better to the date of first documentation of disease progression per RECIST 1.1 and iRECIST respectively.
DOR Assessed by Investigator with iRECIST | Up to 3 years
  DOR is defined as the time from the date of first documentation of a PR/iPR or better to the date of first documentation of disease progression per RECIST 1.1 and iRECIST respectively.
Time to Progression (TTP) Assessed by Investigator with RECIST 1.1 | Up to 3 years
  TTP is defined as the time from the TAK-103 infusion date to the date of first documented disease progression by the investigator per RECIST 1.1 and iRECIST respectively.
TTP Assessed by Investigator with iRECIST | Up to 3 years
  TTP is defined as the time from the TAK-103 infusion date to the date of first documented disease progression by the investigator per RECIST 1.1 and iRECIST respectively.
Progression-Free Survival (PFS) Assessed by Investigator with RECIST 1.1 | Up to 3 years
  PFS is defined as the time from the TAK-103 infusion date to the date of disease progression per RECIST 1.1 and iRECIST respectively or death from any cause, whichever occurs first.
PFS Assessed by Investigator with iRECIST | Up to 3 years
  PFS is defined as the time from the TAK-103 infusion date to the date of disease progression per RECIST 1.1 and iRECIST respectively or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 3 years
  OS is defined as the time from the TAK-103 infusion date to the date of death from any cause.
Cmax: Maximum Observed in Peripheral Blood Drug Concentration after Single Dose Administration by CAR Copy Number | Up to 13 months; Pre-dose and multiple time points (Day 1, 2, 4, 8, 11, 15, 18, 22, 29, Months 3, 4, 5, 7, 10, and 13) post-dose after the intravenous infusion
Tmax : Time of First Occurrence of Maximum Observed Peripheral Blood Concentration by CAR Copy Number | Up to 13 months; Pre-dose and multiple time points (Day 1, 2, 4, 8, 11, 15, 18, 22, 29, Months 3, 4, 5, 7, 10, and 13) post-dose after the intravenous infusion
Clast: Last Observed Quantifiable Concentration in Peripheral Blood by CAR Copy Number | Up to 13 months; Pre-dose and multiple time points (Day 1, 2, 4, 8, 11, 15, 18, 22, 29, Months 3, 4, 5, 7, 10, and 13) post-dose after the intravenous infusion
Tlast: Persistence: Time of Last Observed Quantifiable Concentration in Peripheral Blood (days) by CAR Copy Number | Up to 13 months; Pre-dose and multiple time points (Day 1, 2, 4, 8, 11, 15, 18, 22, 29, Months 3, 4, 5, 7, 10, and 13) post-dose after the intravenous infusion
AUC: Area Under the Blood Concentration-Time Curve by CAR Copy Number | Up to 13 months; Pre-dose and multiple time points (Day 1, 2, 4, 8, 11, 15, 18, 22, 29, Months 3, 4, 5, 7, 10, and 13) post-dose after the intravenous infusion
Number of Participants with Replication Competent Retrovirus (RCR)-Positive Test Results | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/61c2133bf571d4002a64b4bf